CLINICAL TRIAL: NCT04283097
Title: A Phase 1, Multicenter, Open-label, Multiple-ascending Dose Study to Evaluate the Safety, Pharmacokinetics and Clinical Activity of KPG-818 in Subjects With Hematological Malignancies
Brief Title: Safety, Tolerability and Pharmacokinetics Study of KPG-818 in Hematological Malignancies Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kangpu Biopharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KPG-818-HEM-101
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose escalation will use a standard 3+3 approach to establish a maximum tolerated dose (MTD), and the initial escalation dose level will be 2mg/day. Subjects may be enrolled at dose levels 2, 3, 4, and 5 mg and/or intermediate dosing or alternative dosing schedule
Masking Description: This is a open label Phase I study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): KPG-818 dose escalation
  Interventions: Drug: KPG-818

INTERVENTIONS:
Drug: KPG-818 — The 4 planned dose level (cohorts) of KPG-818 will be explored: 2, 3, 4 and 5mg. Each dose of KPG-818 will be administered orally with approximately 240 ml of water daily, and used as a single agent in subjects with selected hematological malignancies (or in combination with dexamethasone weekly for MM), according to specific dosing schedule in each treatment cycle until disease progression, unacceptable toxicity, the subject withdraws, or any other study withdrawal criterion is met. The treatment of study is divided into 6 cycles.
  Other Names: KPG-818 capsules

SUMMARY:
This is a phase 1, multicenter, open-label, multiple-ascending dose study to evaluate the safety, pharmacokinetics and clinical activity of KPG-818 in subjects with hematological malignancies. Approximately 30 patients will be enrolled for dose escalation of 4 dose levels.

Indication: Hematological malignancies (multiple myeloma [MM], mantle cell lymphoma [MCL], diffuse large B-cell lymphoma [DLBCL], adult T-cell leukemia-lymphoma [ATL], and indolent non Hodgkin lymphomas such as follicular lymphoma [FL] and chronic lymphocytic leukemia [CLL]/small lymphocytic lymphoma [SLL]).

DETAILED DESCRIPTION:
This will be a dose escalation study in subjects with selected hematological malignancies. KPG-818 will be used in combination with dexamethasone in subjects with MM, and as monotherapy for other selected hematological malignancies. Each dose of KPG-818 will be administered orally until the completion of treatment cycles, or progressive disease (PD), unacceptable toxicity, the subject withdraws, or any other study withdrawal criterion is met.

The highest dose level which may be tested is 5 mg KPG-818 and dose levels 2, 3, 4, and 5 mg and/or intermediate dosing or alternative dosing schedule may be explored. Each dose level (1-4) will be tested using the standard 3+3 design. DLT will be assessed during the DLT evaluation period (Cycle 1) and the treatment of study is divided into 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Willing and able to provide written consent.
3. Willing and able to adhere to the study visit schedule and other protocol requirements.
4. Hematocytological or pathological diagnosis of MM, MCL, DLBCL, ATL, indolent lymphoma, such as FL and CLL/SLL, etc.
5. Subjects who have relapsed from or are refractory to MM, MCL, DLBCL, ATL, indolent lymphoma, such as FL and CLL/SLL.
6. Have measurable or assessable disease.
7. Meet the laboratory requirements:
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
9. Males and females of childbearing potential must agree to use at least two methods of contraception and continue until 3 months after the completion of study treatment.

Exclusion Criteria:

1. Has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Currently enrolled in another clinical study, except observational studies.
3. Has known active central nervous system metastases and/or lymphomatous meningitis.
4. Persisting toxicities related to prior anticancer treatment > Grade 1.
5. Major surgery or significant traumatic injury within 6 weeks prior to Screening or planned major surgery during the study period.
6. Received live attenuated vaccine within 4 weeks of first dose.
7. Subjects with gastrointestinal disease that may significantly alter the absorption of the study drug.
8. Subjects with a plasma cell leukemia.
9. Subjects with prior history of malignancies, other than MM, lymphoma, or CLL/SLL, unless the subject has been free of the disease for ≥ 5 years.
10. Has a history of anaphylaxis or hypersensitivity to thalidomide, lenalidomide, or pomalidomide.
11. Has known or suspected hypersensitivity to the excipients contained in the formulation of investigational product (IP).
12. Has been treated with an investigational agent (i.e., an agent not commercially available) within 28 days of initiating IP.
13. Prior treatment of any inhibitors of PD-1 or PD-L1 within 3 months prior to initiating IP.
14. Has any one of the following:

    * Clinically significant abnormal ECG finding at Screening.
    * Congestive heart failure.
    * Myocardial infarction within 12 months prior to initiating IP.
    * Unstable or poorly controlled angina pectoris, including the Prinzmetal variant of angina pectoris.
    * Peripheral neuropathy ≥ Grade 2.
    * Subject has taken a strong inhibitor or inducer of CYP3A4/5 including grapefruit, St. John's Wort or related products within 2 weeks prior to dosing and during the course of study.
15. Has current or prior use of immunosuppressive medication within 14 days prior initiating IP.
16. Subject known to test positive for human immunodeficiency virus, active hepatitis B, or active hepatitis C.
17. Subject is unable or unwilling to undergo protocol required thromboembolism prophylaxis.
18. Subject is a female who is pregnant, nursing, or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 6 months of treatment
  Number of Treatment-Emergent Adverse Events(TEAE), serious adverse events (SAEs), dose-limiting toxicities (DLTs), and changes from baseline in laboratory parameters, vital signs, and ECG.
Recommended Phase 2 Dose (RP2D) | Up to 4 weeks of treatment
  Maximum tolerated dose defined as the highest dose level at which 33% or less subjects experience DLT as defined by the protocol.

SECONDARY OUTCOMES:
PK profile of KPG-818: maximum observed plasma concentration (Cmax). | Up to 4 weeks of treatment
PK profile of KPG-818: time of the maximum observed plasma concentration (Tmax) | Up to 4 weeks of treatment
PK profile of KPG-818: area under the plasma concentration-time profile (AUC) from time zero to the last quantifiable concentration (AUC0-t). | Up to 4 weeks of treatment
PK profile of KPG-818: AUC from time zero extrapolated to infinity (AUC0-∞). | Up to 4 weeks of treatment
PK profile of KPG-818: AUC within a dosing interval (AUC0-τ). | Up to 4 weeks of treatment
PK profile of KPG-818: apparent total plasma clearance (CL/F). | Up to 4 weeks of treatment
PK profile of KPG-818: apparent total plasma clearance at steady-state (CLss/F). | Up to 4 weeks of treatment
PK profile of KPG-818: apparent volume of distribution (Vz/F) | Up to 4 weeks of treatment
PK profile of KPG-818: apparent volume of distribution at steady-state (Vss). | Up to 4 weeks of treatment
PK profile of KPG-818: apparent plasma terminal elimination. half-life (t1/2) | Up to 4 weeks of treatment
Assessment of clinical activity: objective response rate (ORR). | Up to 6 months of treatment
  Responses are evaluated based on International Myeloma Working Group (IMWG) Uniform Response Criteria (for MM), Lugano Classification (for lymphoma), International Workshop Group on CLL (iwCLL) Response Criteria, and according to the 'Definition, prognostic factors, treatment, and response criteria of adult T-cell leukemia-lymphoma' (for ATL).
Assessment of clinical activity: disease control rate (DCR). | Up to 6 months of treatment
  Responses are evaluated based on International Myeloma Working Group (IMWG) Uniform Response Criteria (for MM), Lugano Classification (for lymphoma), International Workshop Group on CLL (iwCLL) Response Criteria, and according to the 'Definition, prognostic factors, treatment, and response criteria of adult T-cell leukemia-lymphoma' (for ATL).
Assessment of clinical activity: time to response, duration of response. | Up to 6 months of treatment
  Responses are evaluated based on International Myeloma Working Group (IMWG) Uniform Response Criteria (for MM), Lugano Classification (for lymphoma), International Workshop Group on CLL (iwCLL) Response Criteria, and according to the 'Definition, prognostic factors, treatment, and response criteria of adult T-cell leukemia-lymphoma' (for ATL).
Assessment of clinical activity: progression-free survival. | Up to 6 months of treatment
  Responses are evaluated based on International Myeloma Working Group (IMWG) Uniform Response Criteria (for MM), Lugano Classification (for lymphoma), International Workshop Group on CLL (iwCLL) Response Criteria, and according to the 'Definition, prognostic factors, treatment, and response criteria of adult T-cell leukemia-lymphoma' (for ATL).
Assessment of clinical activity: event-free survival (EFS), and transplantation rate (TR). | Up to 6 months of treatment
  Responses are evaluated based on International Myeloma Working Group (IMWG) Uniform Response Criteria (for MM), Lugano Classification (for lymphoma), International Workshop Group on CLL (iwCLL) Response Criteria, and according to the 'Definition, prognostic factors, treatment, and response criteria of adult T-cell leukemia-lymphoma' (for ATL).

OTHER OUTCOMES:
Biomarkers of KPG-818 | Up to 6 months of treatment
  Aiolos and Ikaros in peripheral blood mononuclear cell (PBMC)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Kangpu Biopharmacuticals
Locations (10):
- United States (10):
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - BRCR Global - USA, Plantation, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - Henry Ford Health System - Hemophilia and Thrombosis Treatment Center, Detroit, Michigan
  - Mohamad Medical Cherry, Morristown, New Jersey
  - Duke University Health System - Duke Endoscopy - Duke Clinic 2H, Durham, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - UPMC CancerCenter, Pittsburgh, Pennsylvania
  - Laguna Clinical Research Associates, Laredo, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No